CLINICAL TRIAL: NCT00807053
Title: A Double-blind, Randomized, Placebo-controlled, Parallel Group, Multicenter, Dose-ranging Study to Assess the Efficacy and Safety of Ciclesonide HFA Nasal Aerosol in Adult and Adolescent Patients 12 Years and Older With Seasonal Allergic Rhinitis (SAR)
Brief Title: Dose-ranging Study to Assess the Efficacy and Safety of Ciclesonide HFA Nasal Aerosol in Adult and Adolescent Patients 12 Years and Older With Seasonal Allergic Rhinitis (SAR) (BY9010/M1-602)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BY9010/M1-602
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-09

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Seasonal Allergic Rhinitis; Ciclesonide; SAR
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Ciclesonide HFA 75 mcg (37,5 mcg / actuation, 1 actuation/nostril), once daily
  Interventions: Drug: Ciclesonide HFA
- 2 (Active Comparator): Ciclesonide HFA 150 mcg (75 mcg / actuation, 1 actuation/nostril), once daily
  Interventions: Drug: Ciclesonide HFA
- 3 (Active Comparator): Ciclesonide HFA 300 mcg (150 mcg / actuation, 1 actuation/nostril), once daily
  Interventions: Drug: Ciclesonide HFA
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide HFA — 75 mcg Ciclesonide HFA versus Placebo
  Arms: 1
Drug: Ciclesonide HFA — 150 mcg Ciclesonide HFA versus Placebo
  Arms: 2
Drug: Ciclesonide HFA — 300 mcg Ciclesonide HFA versus Placebo
  Arms: 3
Drug: Placebo — Placebo
  Arms: 4

SUMMARY:
The primary objective of this study is to demonstrate the efficacy of ciclesonide HFA, applied as a nasal aerosol once daily, in patients with SAR. The secondary objectives are to evaluate Quality-of-Life and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 12 years and older
2. General good health, and free of any concomitant conditions or treatment that could interfere with study conduct,influence the interpretation of study observations/results, or put the patient at increases risk during the trial
3. A history of SAR to relevant seasonal allergen for a minimum of two years immediately preceding the study season. The SAR must have been of sufficient severity to have required treatment (continuous or intermittent) in the past and in the investigator´s judgment - is expected to require treatment throughout the entire study period
4. A demonstrated sensitivity to grass or tree pollen known to induce SAR through a standard skin prick test. A positive test is defined as a wheal diameter at least 3 mm larger than the control wheal for the skin prick test. Documentation of a positive result 12 months prior to screening is acceptable
5. Female is of child-bearing potential and is currently taking and will continue to use a medically reliable method of contraception for the entire study duration (e.g. oral, injectable, trans-cutaneous or implantable contraceptives or intrauterine devices or double-barrier protection). Women of childbearing potential, or less than 1 year postmenopausal, will require a negative pregnancy test at the Screnning Visit (B0) as well as at last on-treatment (T2)
6. Capable of understanding the requirements, risks and benefits of study participation, and, as judged by the investigator, capable of giving informed consent and compliance with all study requirements (visits, record-keeping, etc.)

Exclusion Criteria:

1. Pregnancy, nursing or plans to become pregnant or donate gametes (over a sperm) for in vitro fertilization during the study period or for 30 days following the study period.
2. History of physical findings of nasal pathology, including nasal polyps (within the last 60 days) or other clinically significant respiratory tract malformations, recent nasal biopsy (within the last 60 days), nasal trauma, or surgery and atrophic rhinitis or rhinitis medicamentosa (within the last 60 days)
3. Participation in any investigational drug trial within the 30 days preceding the Screening Visit (B0)
4. A known hypersensitivity to any corticosteroid or any of the excipients in the formulation
5. History of a respiratory infection or disorder (including, but not limited to bronchitis, pneumonia, the common cold, acute or chronic sinusitis, flu, severe acute respiratory syndrome (SARS)) within the 14 days preceding the Screening Visit (B0), or development of a respiratory infection during the Baseline Period.
6. History of alcohol or drug abuse within the preceding two years
7. History of a positive test of HIV, hepatitis B or hepatitis C
8. Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of ß-agonists and any controller drugs (e.g., theophylline, leukotriene antagonists, etc.; intermittent use (less than or equal to 3 uses per week) of inhaled short acting ß-agonists is acceptable
9. Plans to travel outside the study area (the known pollen area for the investigative site) for two or more consecutive days OR 5 or more days total starting from 7 days prior to Randomization Visit (T0) until the final Treatment Visit (T2)
10. Use of any prohibited concomitant medications within the prescribed (per protocol) time since last dose period prior to the Screening Visit (B0) and during entire treatment duration.
11. Use of antibiotic therapy for acute conditions within 14 days prior to the Screening Visit (B0). Low doses of antibiotics taken for prophylaxis are permitted if the therapy was started prior to the Screening Visit (B0) AND is expected to continue throughout the trial.
12. Initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the Screening Visit (B0) AND use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
13. Previous participation in an intranasal ciclesonide HFA nasal aerosol study.
14. Non-vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit (B0).
15. Use of topical corticosteroids in concentrations in excess of 1% hydrocortisone or equivalent within 30 days prior to the Screening Visit (B0); use of a topical hydrocortisone or equivalent in any concentration covering greater than 20% of the body surface; or presence of an underlying condition (as judged by the investigator) that can reasonably be expected to require treatment with such preparations during the course of the study.
16. Initiation of pimecrolimus cream 1% or greater or tacrolimus ointment 0.03% or greater during the study period or planned dose escalation during the study period. However, initiation of these creams/ointments 30 days or more prior to the Screening Visit (B0) AND use of a stable (maintenance) dose during the study period may be considered for inclusion.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2007-04; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Average of AM and PM patient-reported reflective Total Nasal Symptom Score (TNSS) over the first two weeks of treatment | 2 weeks

SECONDARY OUTCOMES:
Average of AM and PM patient-reported instantaneous TNSS over the first two weeks of treatment | 2 weeks
Physician-assessed total nasal symptoms score (PNSS) over the treatment period | 4 weeks
Rhinoconjunctivitis Quality of Life Questionaire (RQLQ) over the treatment period in patients (adolescents and adults) with impaired quality of life at Baseline defined as a RQLQ score of greater than 3.0 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (31):
- United States (31):
  - Altana/Nycomed, Mission Viejo, California
  - Altana/Nycomed, Orange, California
  - Altana/Nycomed, San Diego, California
  - Altana/Nycomed, Colorado Springs, Colorado
  - Altana/Nycomed, Denver, Colorado
  - Altana/Nycomed, Gainsville, Georgia
  - Altana/Nycomed, Savannah, Georgia
  - Altana/Nycomed, Stockbridge, Georgia
  - Altana/Nycomed, Indianapolis, Indiana
  - Altana/Nycomed, Overland Park, Kansas
  - Altana/Nycomed, Bethesda, Maryland
  - Altana/Nycomed, Minneapolis, Minnesota
  - Altana/Nycomed, St Louis, Missouri
  - Altana/Nycomed, Lincoln, Nebraska
  - Altana/Nycomed, Papillion, Nebraska
  - Altana/Nycomed, Skillman, New Jersey
  - Altana/Nycomed, West Brick, New Jersey
  - Altana/Nycomed, Raleigh, North Carolina
  - Altana/Nycomed, Ashland, Oregon
  - Altana/Nycomed, Medford, Oregon
  - Altana/Nycomed, Portland, Oregon
  - Altana/Nycomed, Blue Bell, Pennsylvania
  - Altana/Nycomed, Pittsburgh, Pennsylvania
  - Altana/Nycomed, Upland, Pennsylvania
  - Altana/Nycomed, Charleston, South Carolina
  - Altana/Nycomed, Austin, Texas
  - Altana/Nycomed, New Braunfels, Texas
  - Altana/Nycomed, San Antonio, Texas
  - Altana/Nycomed, Draper, Utah
  - Altana/Nycomed, Burke, Virginia
  - Altana/Nycomed, Richmond, Virginia